CLINICAL TRIAL: NCT03568955
Title: Development and Validation of an Assessment Measure for Prolonged Grief Disorder for Swiss, Japanese and Chinese Bereaved Adults: an Examination of Cultural Differences in Symptoms, Emotion Expression and Regulation
Brief Title: Measurement and Assessment of Prolonged Grief Disorder in Asia
Acronym: MAP Asia
Status: Withdrawn | Type: Observational
Why Stopped: This is no longer considered a clinical trial as per the Kantonial Ethics Committee in Zurich, CH
Sponsor: University of Zurich (Other)
Collaborators: Jichi Medical University (Other); Beijing Normal University (Other)
Responsible Party: Sponsor
Other Study IDs: MAPAsia2018
Record Dates: First submitted 2018-06-01; First posted 2018-06-26 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Prolonged Grief Disorder
Keywords: assessment; validation; prolonged grief disorder; cross cultural; questionnaire
MeSH Terms: conditions — Prolonged Grief Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Swiss Bereaved: Adults from the Swiss population who have lost a loved one at least 6 months to 10 years prior to testing
  Interventions: Diagnostic Test: International Prolonged Grief Disorder Scale (IPGDS)
- Japanese Bereaved: Adults from the Japanese population who have lost a loved one at least 6 months to 10 years prior to testing
  Interventions: Diagnostic Test: International Prolonged Grief Disorder Scale (IPGDS)
- Chinese Bereaved: Adults from the Chinese population who have lost a loved one at least 6 months to 10 years prior to testing
  Interventions: Diagnostic Test: International Prolonged Grief Disorder Scale (IPGDS)

INTERVENTIONS:
Diagnostic Test: International Prolonged Grief Disorder Scale (IPGDS) — Assessment measure for Prolonged Grief disorder based on the ICD-11 (International Classification of Disorders) criteria for PGD (Prolonged Grief Disorder). 15 items

SUMMARY:
The overall project includes three sub-studies. Sub-Study I aims to develop the content of a new cultural sensitive grief questionnaire (International Prolonged Grief Disorder Scale, IPGDS Killikelly and Maercker, 2018) through interviews and focus groups with key (expert) informants and bereaved participants from Japan, Switzerland and China. The content will be piloted in paper and mobile app format. Sub - Study II aims to validate the new paper and mobile questionnaire in 200 participants from each culture using a battery of questionnaires and psychometric assessment. Sub-Study III will explore the relationship between grief and the cultural expression or repression of emotion. This will involve a battery of questionnaires about emotional expression and a short idiographic interview task administered to Swiss, Japanese and Chinese bereaved participants in paper and online format.

DETAILED DESCRIPTION:
Objectives of the project:

The overall aim of this project is to develop three culturally sensitive measures of grief for use in Switzerland, China and Japan. Three sub-aims are described below:

Substudy 1: Development of the questionnaire Substudy 2: Psychometric Validation of the questionnaire Substudy 3: Relationship between emotional expression and grief The relationship between grief and the expression of emotion will be explored within and across the three cultures.

Outcomes of the project:

Sub-study 1:

1. Three new culturally sensitive versions of a Prolonged grief disorder measure (IPGDS) 1) Swiss 2) Japanese 3) Chinese versions: the structure and item content of this measure
2. Beta draft of a mobile app version of the IPGDS questionnaire

   Sub-study 2:
3. Psychometric properties of the IPGDs: specific outcomes including statistical confirmation of the reliability (interrater reliability, test/retest, internal consistency) and validity (criterion, content validity, construct validity) of the IPGDs

   Sub-study 3:
4. Identification and documentation of emotional expression differences in Chinese, Japanese and Swiss culture that may impact on assessment of grief and could inform clinical assessment procedure.

ELIGIBILITY:
Inclusion Criteria:

* Swiss, Japanese, Chinese nationality or identity

  * English, German, Japanese, Cantonese or Mandarin speaking
  * Male and Female subjects 18 years to 75 years of age
  * Written informed consent by the participant after information about the project
  * Loss of a loved one (family or friend) at least 6 months prior, at most 10 years prior

Exclusion Criteria:

* • Severe mental health disorder (e.g. Major depression, suicidality, current schizophrenia),

  * currently in-patient,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be bereaved adult participants from the age of 18 to 65. We will recruit 20 key informants from each country for the qualitative interviews. 150-200 Swiss bereaved, 150-200 Japanese bereaved, 150-200 Chinese bereaved will complete the questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Development and validity of the International Prolonged Grief Disorder Scale (IPGDS), A questionnaire | 24 months
  refinement and psychometric properties of the IPGDS (International Prolonged Grief Disorder Scale): Prolonged grief symptoms will be evaluated through the ICD-11 Prolonged Grief Disorder Scale (IPGDS) (Killikelly and Maercker, 2018). This scale comprises 14 previously used items integrating the PG-13 (Prigerson, Vanderwerker and Maciejewski, 2008) and the SCI-CG (Bui et al., 2015). The participants will be requested to describe how often they had felt preoccupation, yearning and symptoms of emotional distress over the past month because of loss of a loved one, using a 5-point scale: 1 = almost never (less than once a month), 2 = rarely (monthly), 3 = sometimes (weekly), 4 = often (daily), and 5 = always (several times a day). The English, Japanese and Chinese versions of the IPGDs will be translated and back translated following standard protocol (Mollica et al., 1992). The scale will be in paper and online format and can be completed in 5-10 minutes.

SECONDARY OUTCOMES:
Emotional control beliefs about grief scale (ECBG) | 36 months
  Emotion Control Beliefs scale adapted for grief:
  Emotion Control Values on Grief was developed from the existing Emotion Control Values (ECV: Mauss et al., 2010) and adapted to the emotion control of grief. It comprises nine items: (1) "People should not cry a lot when grieving"; (2) "It is helpful to cry a lot when grieving"; (3) "People should not express positive emotions when grieving"; (4) "People should not express negative emotions when grieving"; (5) "It is appropriate to express negative emotions when grieving"; (6) "It is appropriate to express positive emotions when grieving"; (7) "People in general should control their emotions more when grieving"; (8) "It is helpful to express negative emotions when grieving"; (9) "It is helpful to express positive emotions when grieving".
Emotion Regulation Questionnaire (ERQ) | 36 months
  Emotion Regulation Questionnaire The 10-item Emotion Regulation Questionnaire (ERQ) includes two dimensions: cognitive re-appraisal and expression suppression (Gross & Jone, 2003). Each item is rated from from 1 (strongly disagree) to 7 (strongly agree). A higher score indicates a higher frequency to use emotion regulation strategies.
Emotional regulation repertoire(ERR) | 36 months
  Emotion Regulation Repertoire The Emotion Regulation Repertoire (ERR) was developed to assess how close others respond to participants' intense feelings and emotions. For each network member listed in the Social Net-work Index, participants choose from a list of 19 items how the particular network members usually or most often responds to their strong emotions ("This person _____ when I have strong feelings."). Regulation strategies included in the list comprise, amongst others, advises me, understands me, and vents with me. In addition, participants will indicate how their deceased loved one used to re-spond to their emotions.
The social network inventory | 36 months
  Social Network Index The Social Network Index (SNI) was developed and adapted from the existing Social Network Index (SNI: Cohen et al., 1997) in order to tailor it towards social network characteristics of be-reaved individuals. It comprises fourteen items regarding participants' network members including family members, friends, grief support group members, and online contacts. Participants are asked to identify how many network members they feel close to (0-7), and which one of their network members they see or talk to at least once every two weeks (by indicating thei first name and initial for last name).
Idiographic Interview task | 36 months
  Idiographic Interview task (Diminich & Bonanno, 2014) Participants will discuss their relationships with the deceased and current attachment figure in the context of conflict and intimacy will be conducted. Self-reported affect, emotional word use, and facial coding will be measured and compared between groups.
  Participants will be informed that there were no correct answers and that interviewers will be interested in what their particular experiences might be like. Participants will be asked to recall and recount in a fixed order, specific events in which there is: conflict with the deceased; intimacy with the deceased; conflict with other current attachment, and intimacy with other current attachment. The interviewer will halt participant's recounting of the event after 3 minutes.
Positive and Negative Affect Scale | 36 months
  Positive and Negative Affect Scales After each interview topic, participants will be asked to rate using a 5-point Likert scale from 1(very slightly) to 5 (extremely) the extent to which they feel a number of emotions using the Posi-tive and Negative Affect Schedule (PANAS: Watson et al., 1988). The PANAS is composed of two scales, 10 items for positive emotion (interested, excited, strong, enthusiastic, proud, alert, inspired, determined, attentive, active) and 10 items for negative emotion (distressed, upset, guilty, scared, hostile, irritable, ashamed, nervous, jittery, afraid).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Department of Psychopathology and Clinical Intervention, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stelzer EM, Holtge J, Zhou N, Maercker A, Killikelly C. Cross-cultural generalizability of the ICD-11 PGD symptom network: Identification of central symptoms and culturally specific items across German-speaking and Chinese bereaved. Compr Psychiatry. 2020 Nov;103:152211. doi: 10.1016/j.comppsych.2020.152211. Epub 2020 Sep 30. PMID 33049644